CLINICAL TRIAL: NCT03024073
Title: Assessment of Near Vision Capacity in Different Light Intensities and Temperatures in Patients Who Underwent Pseudophakic Presbyopic Correction
Brief Title: Assessment of Near Vision Capacity in Different Light Intensities
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Assistant Professor, Democritus University of Thrace
Other Study IDs: 300/13-1/2017
Record Dates: First submitted 2017-01-14; First posted 2017-01-18 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SG: Study group (patients who underwent pseudophakic presbyopic correction with bilateral bifocal lenses implantation
  Interventions: Procedure: BB-Phaco
- CG: Control group (age-matched participants without pseudophakic presbyopic correction)

INTERVENTIONS:
Procedure: BB-Phaco — Phacoemulsification with bilateral bifocal lenses implantation
  Groups: SG

SUMMARY:
Patients who underwent presbyopic correction with bilateral bifocal intraocular lenses implantation are supposed to have sufficient uncorrected vision capacity for activities of daily living (ADLs) that require near vision acuity (NV), (ie. book reading). However, it is known that light intensity and temperature has a great impact on near vision capacity. Primary objective of this study is to identify the optimal task lighting conditions (in terms of light intensity and temperature) for ADLs that demand near vision acuity for a sample oa patients who underwent presbyopic correction with bilateral bifocal intraocular lenses implantation

ELIGIBILITY:
Inclusion Criteria:

* Presbyopia

Exclusion Criteria:

* Glaucoma
* Corneal pathology
* Fundus pathology
* Severe neurological/mental diseases that interfere with visual acuity

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Presbyopic patients that underwent pseudophakic presbyopic correction with bilateral bifocal intraocular lenses implantation
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01; Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Uncorrected Near Vision Acuity (UnVA) | 6 months
  Near Vision Acuity

SECONDARY OUTCOMES:
Near Vision Capacity (NVC) | 6 months
  NVC score will be measured by the performance score in the following ADLs: a) cellular phone directory entry search, b) reading of message in a cellular phone, c) reading a medical prescription, d) reading a public phonebook

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Principal Investigator — Democritus University of Thrace
Locations (1):
- Democritus University of Thrace, Alexandroupoli, Evros, Greece

IPD SHARING:
Plan to Share IPD: No